CLINICAL TRIAL: NCT05642351
Title: Autobiographical Specificity in Alzheimer's Disease and Behavioral Variant Frontotemporal Dementia
Brief Title: Autobiographical Specificity
Acronym: ESAD
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0626
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Memory; Alzheimer Disease; Frontotemporal Dementia
Keywords: Autobiographical memory; Alzheimer's disease; with behavioral variant of frontotemporal dementia
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alzheimer's Disease: recruited according to criteria by National Institute on Aging (McKhann et al., 2011).
  Interventions: Other: Autobiographical reminder
- Behavioral variant of frontotemporal dementia: recruited following criteria by Rascovsky et al. (2011)
  Interventions: Other: Autobiographical reminder

INTERVENTIONS:
Other: Autobiographical reminder — The analysis of the specificity of Autobiographical Recall will be done through the following scale, developed for the study:
  * 6 points for a recall involving a single personal event located in space AND time (e.g.,"I remember when my parents took me to the sea for the first time..in 1962..in Dunkerque")
  * 5 points for a recall involving a single personal event located in space OR time ("I remember when my parents first took me to the sea...in 1962")
  * 4 points for a recall involving a single personal event but without spatial/temporal details ("I remember when my parents took me to the sea for the first time")
  * 3 points for a recall involving a general personal event but located in space AND time ("we used to go to Dunkerque in the summer")
  * 2 points for a recall involving a general personal event but located in space OR time ("we used to go to Dunkerque")
  * 1 point for a recall involving a general personal event without spatial/temporal details ("we used to go on vacation")

SUMMARY:
Autobiographical memory is diminished in patients with Alzheimer's Disease and those with behavioral variant of frontotemporal dementia, and research has focused on the hampered ability of patients in retrieving specific memories. However, this study proposes a detailed methodology to provide a qualitative analysis of autobiographical specificity.

DETAILED DESCRIPTION:
Patients with Alzheimer's Disease and those with behavioral variant of frontotemporal dementia will be invited to retrieve autobiographical memories. Memories will be analyzed and categorized into specific, categoric, extended, or semantic autobiographical retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer' disease or avioral variant of frontotemporal dementia
* No opposition from the patient to be included in the study
* For Alzheimer's patients: a score of more than 24 out of 30 on the Mini Mental State Examination (McKhann et al., 1984)

Exclusion Criteria:

* Other psychiatric/neurological disorders
* Minor patients
* Adults under guardianship or protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited through the active file of memory consultations of the "memory resource and research center" (CMRR) of the Nantes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Autobiographical specificity | 40 minutes
  We will apply the method by Raes et al. (2007) to assess whether each retrieved event refers to a: specific event, categorical event, extended event, or semantic event

CONTACTS AND LOCATIONS:
Locations (1):
- EL HAJ Mohamad, Nantes, France

IPD SHARING:
Plan to Share IPD: No